CLINICAL TRIAL: NCT03788590
Title: A Prospective, Multicenter, Single-armed Trial That Aims to Evaluate the Safety and Efficacy of Transcatheter Artificial Aortic Valve and Transcatheter Artificial Heart Values Delivery System
Brief Title: Evaluate the Transcatheter Artificial Aortic Valve and Transcatheter Artificial Heart Values Delivery System
Acronym: TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ningbo Jenscare Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT-2017-01
Record Dates: First submitted 2018-12-21; First posted 2018-12-27 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Severe Aortic Stenosis; Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jenscare TAVI (Experimental): Patients undergoing a Jenscare TAVI and delivery system
  Interventions: Device: Jenscare TAVI

INTERVENTIONS:
Device: Jenscare TAVI — Jenscare TAVI and delivery system will implant a percutaneous bioprosthesis value, which is positioned in the native aortic valve, plays a role to control blood flow, and help your heart to work better. It may also shorten your recovery time to getting back to everyday activities.

SUMMARY:
The purpose of this study is to demonstrate that transcatheter artificial aortic valve and transcatheter artificial heart values delivery system is associated with a reduction of all-cause mortality in severe aortic stenosis or insufficiency patients who are high risk or ineligible for aortic valve replacement.

DETAILED DESCRIPTION:
Aortic valve diseases is usually caused by rheumatic fever, congenital aortic valve structural abnormality or degenerative aortic valve calcification. Transcatheter aortic valve implantation (TAVI) has evolved as an alternative to surgical aortic valve replacement (SAVR) with now more than 50,000 implantations in patients with symptomatic severe aortic stenosis, who were considered to be at very high or prohibitive operative risk.

This project take the incidence of all-cause mortality at 12 months since TAVI as the primary endpoint to evaluate the safety and efficacy, then take the procedure success rate, device success rate, incidence of severe adverse events, device operative performance, prosthetic valve performance and quality of life to evaluate transcatheter artificial aortic valve and transcatheter artificial heart values delivery system of Ningbo Jenscare Biotechnology Co., Ltd. in clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 65 years of age;
* Severe aortic stenosis, as defined by ultrasonic cardiogram (peak velocity ≥4.0 m/s, or mean transaortic systolic pressure gradient ≥40 mmHg, or an aortic valve area of <1.0 cm2) or combined merger; severe aortic insufficiency (regurgitation ≥+++ or regurgitation area ≥0.3cm2) combined with left ventricular dilatation ( LVESD≥50mm or LVEDD≥65mm);or severe aortic valve insufficiency combined with left ventricular systolic dysfunction (LVEF<50%);
* Symptoms suggestive of aortic stenosis, NYHA class III or IV;
* Patients who are considered unsuitable for surgery are considered by two or more than two cardiovascular specialists (≥6% using Society of Thoracic Surgeons scoring system estimation; or there is a severe and irreversible organ damage to the patient, such as lung disease, liver disease, kidney disease and so on; or the patient's physical weakness can not be tolerated by surgery; or have other factors affecting surgery, such as postoperative chest radiosurgery, thoracic deformity, and diffuse severe calcification of the aorta, etc);
* A life expectancy of > 1 year;
* Voluntarily participate in and sign the informed consent form and willing to undergo the related examination and clinical follow-up.

Exclusion Criteria:

* Untreated severe coronary stenosis and needs revascularization; or acute myocardial infarction occurred within 1 months, or coronary stent implantation in 1 month;
* Artificial heart valve and artificial valve ring have been implanted；
* Severe mitral insufficiency (regurgitation ≥+++) or mitral stenosis (valvular area<1.5 cm2)；
* left ventricular or atrial thrombus;
* Aortic annulus diameter <17mm or >27 mm;
* Severe left ventricular dysfunction, ejection fraction <20%；
* Severe pulmonary hypertension or severe right ventricular dysfunction；
* The ascending aortic ≥5cm or Aortic root diameter ≥4.5cm;
* Cerebrovascular event in last 3 months；
* Active endocarditis or other active infection;
* Severe renal failure and requires long-term dialysis treatment；
* Severe liver dysfunction；
* Active peptic ulcer；
* Severe coagulation dysfunction; it is known that all anticoagulant schemes are taboo or allergic, or anticoagulants can not be used in the process of testing；
* Severe respiratory failure；
* Severe Alzheimer's disease；
* Patients who were enrolled in any other study in one month;
* Other cases which the researchers believe that it is not suitable to participate in.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2019-02-23 (Estimated); Primary Completion 2021-11-23 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 month
  Cumulative incidence of a combination of all cause death at 12 month after TAVI

SECONDARY OUTCOMES:
Procedure success rate | During the TAVI procedure
  Documentation of no death occurred during or within 72 hours after TAVI, no conversion to conventional cardiopulmonary bypass, the value was placed in the correct anatomical position and achieve the desired effect
Device success rate | During the TAVI procedure
  Documentation of the device was implanted successfully, placed in the correct anatomical position and achieve the desired effect
Incidence of severe adverse events | During the TAVI procedure and 3 days,7 days, 30 days, 3 months, 6 months, 12 months after TAVI
  Documentation of the serious long-term complications, including mortality, stroke, transient ischemic stroke, myocardial infarction, dialysis and reinterventions
Assessment of device operative performance | During the TAVI procedure
  Using the following measure (loading and releasing properties of artificial aortic valve; pushing, emptying, withdrawing, developing performance, fracture of the delivery system) that can be converted to utilities using an algorithm. Utilities range from 1 to 3, with 3 representing perfect performance, and 1 corresponding to the worst performance state.
Echocardiographic assessment of valve performance | 30 days, 3 months, 6 months, 12 months after TAVI
  Using the following measures: effective orifice area (EOA)
Echocardiographic assessment of valve performance | 30 days, 3 months, 6 months, 12 months after TAVI
  Using the following measures: transvalvular mean gradient
Evaluation and improvement of quality of life | Preoperative and 30 days, 3 months, 6 months, 12 months after TAVI
  Measures 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be converted to utilities using an algorithm. Utilities range from 0 to 1, with 1 representing perfect health, and 0 corresponding to the worst imaginable health state.
Echocardiographic assessment of valve performance | 30 days, 3 months, 6 months, 12 months after TAVI
  Using the following measures: peak flow velocity
Echocardiographic assessment of valve performance | 30 days, 3 months, 6 months, 12 months after TAVI
  Using the following measures: degree of aortic valve regurgitation
Echocardiographic assessment of valve performance | 30 days, 3 months, 6 months, 12 months after TAVI
  Using the following measures: degree of perivalvular leakage

CONTACTS AND LOCATIONS:
Overall Officials: Peng Cao, Doctor, Study Director — Ningbo Jenscare Biotechnology Co., Ltd.